CLINICAL TRIAL: NCT01092000
Title: The Nutrition Challenge: A Health Promotion Campaign
Status: Completed | Type: Observational
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Professor, The University of Tennessee, Knoxville
Other Study IDs: IRB: 8087B
Record Dates: First submitted 2010-03-22; First posted 2010-03-24 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Health Promotion; Prevention
Keywords: Health Promotion, Dietary Guidelines, Physical Activity Guidelines
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Faculty/Staff
  Interventions: Behavioral: Monitoring; Other: Education
- Graduate Students
  Interventions: Behavioral: Monitoring; Other: Education
- Undergraduate Students
  Interventions: Behavioral: Monitoring; Other: Education

INTERVENTIONS:
Behavioral: Monitoring — Each week participants are asked to record electronically their fruit intake, vegetable intake and minutes of physical activity.
Other: Education — Monthly exercise tips handout.

SUMMARY:
The purpose of the challenge is to see if we, as the nutrition experts, can follow the dietary and physical activity guidelines promoted to the public. We have an opportunity to "practice what we preach." Scientific evidence demonstrates, knowledge is not enough to change ones'behaviors. It is through positive approaches and lifestyle changes that behavior can be altered. By experiencing the planning, work, and motivation required to make lifestyle changes we can all be better clinicians.

ELIGIBILITY:
Inclusion Criteria:

* Regular access to the internet

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All participants in each group are associated with the Department of Nutrition at the Unviersity of Tennessee.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Average Cups of Fruit per Day | 12-weeks
Average Cups of Vegetables per Day | 12 weeks
Average Minutes of Physical Activity Per Week | 12-weeks

CONTACTS AND LOCATIONS:
Overall Officials: Susan B MacArthur, Principal Investigator — Healthy Eating and Activity Laboratory, University of Tennessee; Shannon M Looney, MS, MPH, Study Chair — Healthy Eating and Activity Laboratory, University of Tennessee; Hollie A Raynor, PhD, RD, LDN, Study Director — Faculty Advisor: Assistant Professor
Locations (1):
- The Department of Nutrition at the University of Tennessee, Knoxville, Knoxville, Tennessee, United States